CLINICAL TRIAL: NCT00314158
Title: A Study of a Glaucoma Therapy to Treat Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-05-24
Record Dates: First submitted 2006-04-10; First posted 2006-04-13 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2012-03

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — brinzolamide; Timolol; Ophthalmic Solutions; Suspensions; Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Brinzolamide +Timolol (Experimental)
  Interventions: Drug: Brinzolamide 10 mg/ml + Timolol 5 mg/ml eye drops, suspension
- Brinzolamide (Active Comparator)
  Interventions: Drug: Brinzolamide 10 mg/ml (AZOPT) eye drops, suspension
- Timolol (Active Comparator)
  Interventions: Drug: Timolol 5 mg/ml eye drops, solution

INTERVENTIONS:
Drug: Brinzolamide 10 mg/ml + Timolol 5 mg/ml eye drops, suspension — One drop twice daily in each study eye for six months
  Arms: Brinzolamide +Timolol
Drug: Brinzolamide 10 mg/ml (AZOPT) eye drops, suspension — One drop twice daily in each study eye for six months
  Other Names: AZOPT
  Arms: Brinzolamide
Drug: Timolol 5 mg/ml eye drops, solution — One drop twice daily in each study eye for six months
  Arms: Timolol

SUMMARY:
The purpose of this study is to determine whether a glaucoma therapy is safe and effective in treating patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of open-angle glaucoma
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Under 18
* Pregnant
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 523 (Actual)
Dates: Start 2005-11; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Mean intra-ocular pressure (IOP)

CONTACTS AND LOCATIONS:
Locations (1):
- United States Investigative Sites, Fort Worth, Texas, United States

REFERENCES:
- [Result] Kaback M, Scoper SV, Arzeno G, James JE, Hua SY, Salem C, Dickerson JE, Landry TA, Bergamini MV; Brinzolamide 1%/Timolol 0.5% Study Group. Intraocular pressure-lowering efficacy of brinzolamide 1%/timolol 0.5% fixed combination compared with brinzolamide 1% and timolol 0.5%. Ophthalmology. 2008 Oct;115(10):1728-34, 1734.e1-2. doi: 10.1016/j.ophtha.2008.04.011. Epub 2008 Jun 5. PMID 18538406